CLINICAL TRIAL: NCT03468322
Title: A Double-blind, Intra-individual Comparison, Proof-of-concept Trial of Topical AC-203 in Patients With Inherited Epidermolysis Bullosa
Brief Title: A Double-blind, Intra-individual Comparison, POC Trial of AC-203 in EB Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-203-EBS-005
Record Dates: First submitted 2018-03-08; First posted 2018-03-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Inherited Epidermolysis Bullosa
MeSH Terms: interventions — diacerein

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AC-203 1% ointment (Experimental): AC-203 1% ointment, QD
  Interventions: Drug: AC-203
- Vehicle ointment (Placebo Comparator): Vehicle ointment, QD
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AC-203 — The investigational product is formulated as 1% topical ointment
  Arms: AC-203 1% ointment
Drug: Vehicle — Vehicle-only control study medication is the same formulation as investigational product without active ingredient
  Arms: Vehicle ointment

SUMMARY:
Inherited epidermolysis bullosa (EB) is a genetic skin disorder characterized by skin fragility and recurrent blister formation. More and more evidence has suggested that the skin lesions initially caused by genetic mutations may be further aggravated by inflammatory responses. Several reports showed successful alleviation of EB symptoms upon treatment with immunomodulatory therapies. Modulation of proinflammatory cytokine IL-1β has shown promising results in alleviating epidermolysis bullosa simplex (EBS), a major subtype of inherited EB, by downregulating IL-1β-mediated JNK/MAPK signaling pathway. This data further supports the potential of using cytokine modulators to treat EB.

AC-203, a topical formulation, can inhibit the production and activity of IL-1β, down-regulate IL-1β receptors, and increase IL1β-receptor antagonist (IL1-Ra) expression. In addition, AC-203 has been reported to inhibit anti-BP180 autoantibody-induced IL-6/IL-8 upregulation in cultured keratinocytes and LPS-induced IL-6 upregulation in cultured macrophages. Furthermore, AC-203 was also found to inhibit the formation of NLRP3 inflammasome, which plays essential roles in induction of caspase-1-dependent pyroptosis and release of inflammatory cytokines IL-1β and IL-18. These studies demonstrated the cytokine modulatory properties of AC-203 and pointed out the possible application of AC-203 in a variety of inflammatory diseases.

This study is designed to test the efficacy, safety, tolerability, and pharmacokinetics of AC-203 ointment (vs. placebo) in patients with inherited EB.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 2 years of age.
2. Subject has a clinical diagnosis of EB.
3. Subject has a laboratory confirmed diagnosis of inherited EB based on electron microscopy and/or immunofluorescence antigenic mapping.
4. Subject has two comparable areas with 1% - 5% BSA each. These two areas could be on any body surface except the face, scalp, groin, palms and soles. Percentage BSA of the designated areas within subject should be the same. Comparable areas are defined as having similar lesion (i.e., blisters, erosions, erythema and crusts) history and current lesion status by investigator's judgement on each area at Screening Visit (Visit 1) and Day 1 (Visit 2).
5. Is male, or is female and meets all the following criteria:

   1. Not breastfeeding
   2. If of childbearing potential (defined as non-post-hysterectomy or non-post-menopausal [≥50 years of age and amenorrheic for at least 1 year]), must have a negative pregnancy test result at Visit 1, and must practice and be willing to continue to practice appropriate birth control during the entire duration of the study.
6. Is able to read, understand, and sign the Informed Consent Form (ICF), answer the study questionnaires, communicate with the investigator, and understand and comply with protocol requirements, OR Informed consent received from subject's parents/caregiver or legal guardian (when subject < 20 years).

Exclusion Criteria:

1. Subject has a current malignancy, or a history of treatment for a malignancy within two years.
2. Systemic infections.
3. Subjects who are pregnant, lactating, or planning a pregnancy during the study.
4. History of allergy or hypersensitivity to any component of study medication.
5. Any other significant diseases, conditions, or laboratory values which, in the opinion of the investigator, might make participation not in the subject's best interest or confound the interpretation of study results.
6. Any prior use of approved or investigational biologic anti-inflammatory therapy within 6 months prior to screening, including but not limited to: anakinra, rilonacept, canakinumab, etanercept, adalimumab, infliximab, rituximab, certolizumab, golimumab, tocilizumab, bertilimumab, or abatacept.
7. Use of non-steroid immunosuppressants including but not limited to azathioprine, mycophenolate, cyclophosphamide, chlorambucil, methotrexate, tacrolimus, or cyclosporine in the 2 weeks prior to screening.
8. Has been treated with gentamicin within 90 days prior to screening (Note: products containing gentamicin used on eyes are allowed).
9. Has been treated with minocycline, oxytetracycline, tetracycline or doxycycline within 7 days prior to screening.
10. Subjects has used any topical allantoin ≥ 3% within 30 days prior to screening.
11. Has been treated systemic steroid within 30 days prior to screening.
12. Prior treatment with any investigational therapy within 30 days prior to screening.
13. Is an immediate family member (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study at the clinical study site, or is directly affiliated with the study at the clinical study site.
14. Is employed by sponsor (i.e., is an employee, temporary contract worker, or designee responsible for the conduct of the study).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Percentage change in lesion surface area from baseline by treatment | 2, 4, 5, 6, 8, 12 Weeks

SECONDARY OUTCOMES:
Percentage change in blister number from baseline by treatment | 2, 4, 5, 6, 8, 12 Weeks
Proportion of subjects with at least 40% reduction in blister number from baseline by treatment | 2, 4, 5, 6, 8, 12 Weeks
Pruritus assessment scale changes from baseline by treatment | 2, 4, 5, 6, 8, 12 Week
  100-mm line (anchored at 0 mm for no pruritus, 100 mm for worst possible pruritus)
Pain assessment scale changes from baseline by treatment | 2, 4, 5, 6, 8, 12 Weeks
  100-mm line (anchored at 0 mm for no pruritus, 100 mm for worst possible pruritus)
IL-1beta concentrations and changes from baseline | 8 Weeks
hsCRP concentrations and changes from baseline | 8 Weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Mackay Memorial Hospital, Hsinchu
  - National Cheng Kung University Hospital, Tainan